CLINICAL TRIAL: NCT06148636
Title: A Phase 1, First-in-human Clinical Trial of [212Pb] VMT-alpha-NET Using a Forward Dosimetric Planning Technique to Treat Refractory or Relapsed Neuroendocrine Tumors
Brief Title: A Safety Study of 212Pb-VMT-alpha-NET in Patients With Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: David Bushnell (Other)
Collaborators: Holden Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH); Perspective Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, David Bushnell, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202206110; R01CA243014 (NIH)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Tumor of the Lung; Neuroendocrine Tumor Grade 1; Neuroendocrine Tumor Grade 2; Neuroendocrine Tumor of Pancreas
Keywords: alpha therapy; recurrent disease; theranostics; nuclear medicine
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell; Recurrence

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- -1 Dose Level (Experimental): This dose level is used if the starting dose level is deemed to have unacceptable toxicity.
  Participants are prescribed [212Pb] VMT-α-NET with the total radiation dose to kidneys not to exceed 200 cGy.
  Interventions: Drug: [212Pb] VMT-α-NET; Diagnostic Test: [203Pb] VMT-α-NET SPECT/CT
- Cohort 1 (Experimental): This is the starting dose level for participants. Participants are prescribed [212Pb] VMT-α-NET with the total radiation dose to kidneys not to exceed 350 cGy.
  Interventions: Drug: [212Pb] VMT-α-NET; Diagnostic Test: [203Pb] VMT-α-NET SPECT/CT
- Cohort 2 (Experimental): If the participants from Cohort 1 tolerate therapy, new participants are enrolled and are prescribed [212Pb] VMT-α-NET with the total radiation dose to kidneys not to exceed 600 cGy.
  Interventions: Drug: [212Pb] VMT-α-NET; Diagnostic Test: [203Pb] VMT-α-NET SPECT/CT
- Cohort 3 (Experimental): If the participants from Cohort 2 tolerate therapy, new participants are enrolled and are prescribed [212Pb] VMT-α-NET with the total radiation dose to kidneys not to exceed 810 cGy.
  Interventions: Drug: [212Pb] VMT-α-NET; Diagnostic Test: [203Pb] VMT-α-NET SPECT/CT
- Cohort 4 (Experimental): If the participants from Cohort 3 tolerate therapy, new participants are enrolled and are prescribed [212Pb] VMT-α-NET with the total radiation dose to kidneys not to exceed 1050 cGy.
  Interventions: Drug: [212Pb] VMT-α-NET; Diagnostic Test: [203Pb] VMT-α-NET SPECT/CT

INTERVENTIONS:
Drug: [212Pb] VMT-α-NET — Up to 2 infusions with [212Pb] VMT-α-NET, each infusion separated by at least 8 weeks. During each infusion, the participants also receive an infusion with lysine and arginine (amino acids) to help reduce kidney damage.
Diagnostic Test: [203Pb] VMT-α-NET SPECT/CT — The [203Pb] VMT-α-NET SPECT/CT is performed for all participants to determine trial eligibility as well as for the calculations to determine the estimated radiation dose to kidneys. This involves three imaging sessions of about 2 hours each over 2 days. The participants also receive an infusion with lysine and arginine (amino acids) to help reduce kidney damage at the time they receive the injection of . [203Pb] VMT-α-NET, a radioactive tracer drug.

SUMMARY:
This is a safety study to determine the recommended dose to test in clinical trials. The study involves two treatments with 212Pb (212-lead) VMT-α-NET. This is a safety study only; it will most likely not provide therapeutic benefit.

DETAILED DESCRIPTION:
This research study is designed to explore if a new radiotherapeutic (radioactive) drug, named 212Pb (212-lead) VMT-α-NET, works against neuroendocrine tumor cells. To begin researching this drug, we need to determine if [212Pb] VMT-α-NET is safe and tolerable when used as a cancer treatment. As a safety study, it is unknown if the treatment is safe or effective.

The study will also estimate the radiation dose to the kidneys for this treatment. To calculate this radiation dose, imaging is also performed with the sister drug, [203Pb] VMT-α-NET using SPECT/CT imaging. Each participant is assigned a radiation dose to the kidneys that cannot be exceeded. The study is testing the safety of the specific radiation dose to the kidneys when using [212Pb] VMT-α-NET.

Participants are assigned a radiation dose based on how other participants have tolerated the [212Pb] VMT-α-NET. The amount of [212Pb] VMT-α-NET administered varies person-to-person because of each person's unique tumor uptake of [203Pb] VMT-α-NET and how long it lasts in the body.

The study involves 2 treatments, about 8 to 10 weeks apart. The drug is given by infusion once per treatment. The participants also receive an infusion of amino acids to help protect the kidneys as well as medications to help protect against nausea (feeling sick to the stomach).

Once a participant is administered the [212Pb] VMT-α-NET, they must be followed (i.e. come back to the clinic) for at least 6 months for safety assessments. Safety assessments include blood tests to check bone marrow, kidney, and liver function as well as urinary tests to check kidney function. Participants will also have imaging at 6 months post-treatment to measure how their tumors responded to therapy.

Participants will have lifelong follow-up for this study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to provide informed consent
* Stated willingness to comply with all study procedures and availability for duration of study
* Aged ≥ 18 years to 80 years at the time of study drug administration
* Pathologically confirmed (histology or cytology) malignant neoplasm that is determined to be a well-differentiated neuroendocrine tumor (i.e. grade 1 or grade 2)
* Disease not amenable to curative intent treatment (e.g., surgery) and in addition, has shown either clinical or radiographic progression on all available therapies known to confer clinical benefit in the opinion of the referring physician. If a patient is suspected of experiencing a clinical non-response to current treatment (i.e., the patients clinical symptomatology has not improved despite treatment) the patient may be included if confirmed by the study investigator.
* Prior peptide receptor radionuclide therapy (PRRT)
* Positive somatostatin receptor (SSTR) PET/CT utilizing an FDA approved agent within 12 months prior to anticipated day 1 of treatment demonstrating SSTR positive tumor sites.
* ≥1 evaluable site of disease measuring ≥ 1.0 cm in diameter on CT or MRI as measured per RECIST
* Adequate performance status (ECOG of 0 or 1; or KPS of ≥70).
* No other active malignancy that requires immediate treatment. Slow growing concurrent cancers (such as prostate cancer) are acceptable with appropriate documentation from their treating oncologists for that primary.
* Not experiencing an uncontrolled intercurrent illness such as: infection requiring inpatient admission, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations, or any other condition that would limit compliance with study requirements as determined by study team members.
* Agreement to adhere to Lifestyle Considerations throughout study duration:

During this study, participants are asked to:

* Refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice, [pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices] from the day prior to therapy through 5 days post-treatment.
* Comply with their antihypertensive medications, if prescribed.
* Refrain from excessive alcohol use.
* Refrain from "natural" or "herbal" supplements unless approved by the treating physician and research team.
* Utilize contraception for at least 6 months in uterine-bearing patients and at least 3 months in testes-bearing patients.

Exclusion Criteria:

* Platelets < 100,000 k/mm3
* Absolute neutrophil count (ANC) of < 1500 cells/mm3
* Total bilirubin ≥ 2.5x institutional upper limit of normal for age and weight
* Aspartate aminotransferase (AST) > 2.5 x the institutional upper limit of normal
* Alanine aminotransferase (ALT)> 2.5 x the institutional upper limit of normal
* eGFR < 50 mL/min/1.73 m2 (using the Cockcroft Gault formula)
* Proteinuria grade 2 (i.e., ≥ 3+ proteinuria)
* Individuals who are pregnant or breast feeding. A pregnancy test will be administered to individuals of child-bearing potential (per institutional policies) at screening. Participants must agree to pregnancy tests prior to each administration of a radionuclidic agent for this study.
* Individuals of reproductive potential who decline to use effective contraception through the study. Contraception should only be stopped after a conversation with the attending oncologist.
* Lactating individuals who decline to withhold breastfeeding their child. Participants may not breast feed during this study and should only resume after the study in consultation with their oncologist.
* Patient with increased fall risk in the opinion of healthcare professionals
* Therapy (including radiation therapy) within 2 calendar weeks of the start of study therapy. (Toxicities from prior therapies should have resolved to ≤ CTCAE grade 1 or a new baseline established).
* Therapeutic investigational drug within 4 weeks of C1D1 (imaging agents are acceptable)
* History of congestive heart failure and cardiac ejection fraction ≤ 40%
* Patients for whom, in the opinion of their physician, a 24-hour discontinuation of somatostatin analogue therapy represents a health risk.
* Long-acting somatostatin analogue treatment ≤ 14 days of C1D1
* Prior external beam radiation dose of >16 Gy to the kidneys.
* Prior external beam radiation (including brachytherapy) involving 25% of the bone marrow (excluding scatter doses of ≤ 5 Gy) as estimated by a radiation oncologist.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 90Y-DOTA-tyr3-Octreotide, Octreoscan®, or 68Ga-Octreotide.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine recommended therapeutic dose of [212Pb] VMT-α-NET | From study day 1 through 6 months post-treatment
  Determine the recommended phase 2 dose for therapy with [212Pb]VMT-Α-NET administered intravenously to patients with neuroendocrine tumors that have progressed despite therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At 6 months post-treatment
  Determine objective response rate using the standardized technique (RECISTv1.1) in patients with treatment refractory neuroendocrine tumors (NETs) when treated with [212Pb] VMT-α-NET. Objective response rate is the incidence of complete response and partial response added together.
Maximum tolerated radiation dose for kidneys | From study day 1 through 12 months post treatment
  Determine the maximum tolerated critical organ dose limit for kidneys for therapy with [212Pb]VMT-α-NET administered intravenously to patients with neuroendocrine tumors that have progressed despite therapy.
  Maximum tolerated radiation dose is indicated by the number and severity of renal (i.e. kidney) toxicities observed through 12 months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Bushnell, MD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center at the University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
A HIPAA limited dataset will be shared with requestors for each participant who has provided consent to data sharing. Data will represent critical and / or key data for primary and secondary objectives. Codebook defining data, as well as the protocol, consent, and statistical analysis plan will also be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of study.
Access Criteria: Data Usage Agreement (DUA) must be executed between University of Iowa and requestor/requestor's organization.